CLINICAL TRIAL: NCT00814710
Title: Primary Vaccination Course in Healthy Children Receiving the Pneumococcal Vaccine GSK 1024850A Co-administered With Tritanrix™-HepB/Hib at 6, 10 and 14 Weeks of Age
Brief Title: Primary Vaccination Study With a Pneumococcal Conjugate Vaccine in Healthy Children 6 to 10 Weeks of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 111188; 2011-004644-22 (EudraCT Number)
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae
Keywords: Pneumococcal disease; Pneumococcal vaccine; Safety; Primary vaccination; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — Hiberix; Tritanrix-HepB vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Synflorix & Tritanrix-HebB/Hib Group (Experimental): Subjects received SynflorixTM (GSK1024850A) intramuscularly in the right thigh co-administered with TritanrixTM-HepB/Hib intramuscularly in the left thigh at 6-10-14 weeks of age (=study month 0, 1, 2)
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib
- Hiberix group & Tritanrix-HebB Group (Active Comparator): Subjects received HiberixTM intramuscularly in the right thigh co-administered with TritanrixTM-HepB intramuscularly in the left thigh at 6-10-14 weeks of age (=study month 0, 1, 2)
  Interventions: Biological: Hiberix; Biological: Tritanrix-HepB

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 3 doses
  Arms: Synflorix & Tritanrix-HebB/Hib Group
Biological: Tritanrix-HepB/Hib — Intramuscular injection, 3 doses
  Other Names: DTPw-HBV/Hib
  Arms: Synflorix & Tritanrix-HebB/Hib Group
Biological: Hiberix — Intramuscular injection, 3 doses
  Other Names: Hib
  Arms: Hiberix group & Tritanrix-HebB Group
Biological: Tritanrix-HepB — Intramuscular injection, 3 doses
  Other Names: DTPw-HBV
  Arms: Hiberix group & Tritanrix-HebB Group

SUMMARY:
The purpose of this study is to assess the immunogenicity in terms of antibody response and the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following primary vaccination of Indian infants with pneumococcal conjugate vaccine GSK1024850A co-administered with a diphtheria, tetanus, whole cell pertussis (DTPw)-combined vaccine during the first 4 months of life. The study will be conducted in India.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-10 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol.
* Written or oral, signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child/ward. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Free of any known or suspected health problems (as established by medical history and clinical examination before entering into the study).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (with the exception of hepatitis B immunoglobulins at birth).
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae (with the exception of hepatitis B vaccination at birth or at least 30 days before the subject's first study visit).
* History of, or intercurrent, diphtheria, tetanus, pertussis, hepatitis B, Streptococcus and Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Babies for which birth weight is < 2 kilogram.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2009-03-07 (Actual); Primary Completion 2009-11-13 (Actual); Study Completion 2009-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- India (4):
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vellore

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=260

REFERENCES:
- [Background] Lalwani S, Chatterjee S, Chhatwal J, Verghese VP, Mehta S, Shafi F, Borys D, Moreira M, Schuerman L. Immunogenicity, safety, and reactogenicity of the 10-valent pneumococcal non-typeable Hemophilus influenzae protein D conjugate vaccine (PHiD-CV) when co-administered with the DTPw-HBV/Hib vaccine in Indian infants: a single-blind, randomized, controlled study. Hum Vaccin Immunother. 2012 May;8(5):612-22. doi: 10.4161/hv.19287. Epub 2012 May 1. PMID 22634448
- [Derived] Lalwani S, Chatterjee S, Chhatwal J, Simon A, Ravula S, Francois N, Mehta S, Strezova A, Borys D. Randomized, open-label study of the impact of age on booster responses to the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in children in India. Clin Vaccine Immunol. 2014 Sep;21(9):1292-300. doi: 10.1128/CVI.00068-14. Epub 2014 Jul 9. PMID 25008901
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111188 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Synflorix and Tritanrix-HepB/Hib Group: Subjects received SynflorixTM (GSK1024850A) intramuscularly in the right thigh co-administered with TritanrixTM-HepB/Hib intramuscularly in the left thigh at 6-10-14 weeks of age (=study month 0, 1, 2)
- Hiberix Group and Tritanrix-HepB Group: Subjects received HiberixTM intramuscularly in the right thigh co-administered with TritanrixTM-HepB intramuscularly in the left thigh at 6-10-14 weeks of age (=study month 0, 1, 2)
Period: Overall Study
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Started | 240 | 120
Completed | 232 | 117
Not Completed | 8 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group | Total
Number analyzed (Participants) | 240 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.7 (1.08) | 6.7 (1.05) | 6.7 (1.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 66 | 175
  Male | 131 | 54 | 185

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes
Description: Concentrations were expressed as Geometric Mean Concentrations (GMCs) in microgram per milliliter (µg/mL).
  Pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after primary immunization (month 3)
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects with available immunogenicity data.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 229 | 116
µg/mL
  Anti-1 | 3.27 [2.91 to 3.67] | 0.03 [0.03 to 0.04]
  Anti-4 | 3.80 [3.33 to 4.33] | 0.04 [0.03 to 0.05]
  Anti-5 | 4.17 [3.72 to 4.67] | 0.05 [0.04 to 0.05]
  Anti-6B | 0.71 [0.59 to 0.86] | 0.05 [0.04 to 0.06]
  Anti-7F | 3.87 [3.47 to 4.31] | 0.06 [0.05 to 0.07]
  Anti-9V | 4.21 [3.71 to 4.78] | 0.06 [0.05 to 0.08]
  Anti-14 | 5.21 [4.51 to 6.01] | 0.26 [0.20 to 0.34]
  Anti-18C | 15.23 [12.96 to 17.90] | 0.07 [0.05 to 0.08]
  Anti-19F | 11.78 [10.26 to 13.53] | 0.12 [0.10 to 0.16]
  Anti-23F | 1.18 [0.98 to 1.42] | 0.05 [0.04 to 0.05]

2. Primary Outcome: Concentration of Antibody Against Protein D (PD)
Description: Concentrations were expressed as GMCs GSK's 22F-inhibition in enzyme-linked-immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 227 | 116
EL.U/mL | 2981.7 [2703.0 to 3289.2] | 63.9 [55.8 to 73.1]

3. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Pneumococcal Serotypes
Description: Vaccine pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
  Cross-reactive pneumococcal serotypes included 6A and 19A.
  Opsonophagocytic activity was defined as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay was an opsonic titer equal to or greater than 8.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 116 | 57
subjects
  Opsono-1 (N=116; 57) | 105 | 3
  Opsono-4 (N=116; 55) | 114 | 24
  Opsono-5 (N= 116; 56) | 111 | 2
  Opsono-6B (N=116; 54) | 98 | 5
  Opsono-7F (N=116; 53) | 116 | 35
  Opsono-9V (N=115; 56) | 113 | 9
  Opsono-14 (N=115; 56) | 110 | 14
  Opsono-18C (N=115; 55) | 113 | 2
  Opsono-19F (N=116; 56) | 114 | 7
  Opsono-23F (N=116; 54) | 113 | 9
  Opsono-6A (N=110;57) | 54 | 7
  Opsono-19A (N=109;57) | 35 | 0

4. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Serotypes Equal to or Above Cut-off Value
Description: Vaccine pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Cross-reactive pneumococcal serotypes included 6A and 19A.
  The cut-off was defined as 0.20 microgram per milliliter (µg/mL).
Time Frame: One month after primary immunization
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 229 | 116
subjects
  Anti-1 | 228 | 2
  Anti-4 | 225 | 10
  Anti-5 | 226 | 10
  Anti-6B | 178 | 9
  Anti-7F | 228 | 16
  Anti-9V | 227 | 21
  Anti-14 | 229 | 66
  Anti-18C | 227 | 20
  Anti-19F | 227 | 40
  Anti-23F | 205 | 12
  Anti-6A (N=229;115) | 95 | 12
  Anti-19A | 146 | 21

5. Secondary Outcome: Concentrations of Antibodies Against Pneumococcal Cross-reactive Serotypes
Description: Concentrations were expressed as GMCs in µg/mL. Pneumococcal cross-reactive serotypes included 6A and 19A.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 229 | 116
µg/mL
  Anti-6A (N=229;115) | 0.15 [0.13 to 0.18] | 0.06 [0.05 to 0.08]
  Anti-19A | 0.33 [0.27 to 0.39] | 0.08 [0.06 to 0.09]

6. Secondary Outcome: Number of Subjects Seropositive for Pneumococcal Serotypes
Description: Vaccine pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Cross-reactive pneumococcal serotypes included 6A and 19A.
  Seropositivity was defined as a titer equal to or greater than 0.05 µg/mL
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 229 | 116
subjects
  Anti-1 | 228 | 19
  Anti-4 | 228 | 24
  Anti-5 | 229 | 46
  Anti-6B | 215 | 40
  Anti-7F | 229 | 52
  Anti-9V | 228 | 49
  Anti-14 | 229 | 101
  Anti-18C | 227 | 56
  Anti-19F | 229 | 90
  Anti-23F | 220 | 37
  Anti-6A (N=229;115) | 188 | 62
  Anti-19A | 207 | 71

7. Secondary Outcome: Number of Subjects Seropositive for Protein D (PD)
Description: Seropositivity for PD was defined greater than or equal to 100 EL.U/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 227 | 116
subjects | 226 | 16

8. Secondary Outcome: Concentration of Antibody Against Polyribosyl-ribitol Phosphate (PRP)
Description: Concentration is expressed as GMC in µg/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
µg/mL | 31.367 [26.417 to 37.246] | 34.415 [26.847 to 44.116]

9. Secondary Outcome: Concentration of Antibodies Against Diphteria (Anti-DT) and Tetanus (Anti-TT)
Description: Concentrations were expressed as GMCs in international units per milliliter (IU/mL).
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
IU/mL
  Anti-DT | 2.580 [2.146 to 3.102] | 2.065 [1.736 to 2.457]
  Anti-TT | 3.726 [3.182 to 4.363] | 1.542 [1.316 to 1.807]

10. Secondary Outcome: Concentration of Antibody Against Bordetella Pertussis (B. Pertussis)
Description: Concentration was expressed as GMC in EL.U/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
EL.U/mL | 90.3 [80.3 to 101.6] | 114.5 [101.2 to 129.5]

11. Secondary Outcome: Concentration of Antibody Against Hepatitis B (Anti-HBs) by Enzyme-Linked ImmunoSorbent Assay (ELISA).
Description: Concentration was expressed as GMC in milli international units per milliliter (mIU/mL). As a decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL), the table shows results following partial or complete retesting/reanalysis.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 92 | 89
mIU/mL | 1970.5 [1614.9 to 2404.5] | 1378.2 [1115.6 to 1702.6]

12. Secondary Outcome: Number of Subjects Seropostive for B. Pertussis
Description: Seropositivity was defined as and antibody concentration equal to or greater than 15 EL.U/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
subjects | 113 | 116

13. Secondary Outcome: Number of Seroprotected Subjects (Anti-DT, Anti-TT, Anti-PRP, Anti-HBs)
Description: Seroprotection was defined as:
  Anti-DT antibody concentration equal to or greater than 0.1 IU/mL. Anti-TT antibody concentration equal to or greater than 0.1 IU/mL. Anti-PRP antibody concentration equal to or greater than 0.15 µg/mL Anti-HBs antibody concentration greater than or equal to 10 mIU/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
subjects
  Anti-DT | 113 | 116
  Anti-TT | 113 | 116
  Anti-PRP 0.15 | 113 | 115
  Anti-HBs (N=92,89) | 92 | 89

14. Secondary Outcome: Number of Seroprotected Subjects (Anti-PRP Above the Cut-off of 1.0 µg/mL)
Description: Anti-PRP antibody concentration equal to or greater than 1.0 µg/mL.
Time Frame: One month after primary immunization (month 3)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 113 | 116
subjects | 113 | 114

15. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms
Description: Solicited local symptoms included pain, redness and swelling. Solicited general symptoms included drowsiness, fever (equal to or above 38 degrees Celsius and above 39 degrees Celsius), irritability and loss of appetite.
Time Frame: Within 4 days (day 0-3) after vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects. However, the total number of subjects analyzed in this Total Vaccinated cohort included all subjects having returned their symptom sheets.
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 238 | 119
subjects
  Pain | 209 | 105
  Redness | 128 | 76
  Swelling | 166 | 83
  Drowsiness | 73 | 34
  Fever ≥38.0˚C | 182 | 85
  Fever >39.0˚C | 24 | 5
  Irritability | 178 | 88
  Loss of appetite | 96 | 49

16. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms
Time Frame: Within 31 days (day 0-30) after vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 240 | 120
subjects | 38 | 17

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Following first vaccination (Month 0) throughout the entire study period (month 3)
Population: Analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Number analyzed (Participants) | 240 | 120
subjects | 5 | 1

ADVERSE EVENTS:
Time Frame: For other AEs day 0-3 (solicited) and day 0-30 unsolcited. For SAEs month 0 to Month 3.
Arm/Group | Synflorix and Tritanrix-HepB/Hib Group | Hiberix Group and Tritanrix-HepB Group
Serious Adverse Events (participants affected / at risk) | 5/240 | 1/120
Other Adverse Events (participants affected / at risk) | 231/240 | 114/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix and Tritanrix-HepB/Hib Group (N=240) | Hiberix Group and Tritanrix-HepB Group (N=120)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Bronchopneumonia (Infections and infestations) | 2 | 1
Chikungunya virus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix and Tritanrix-HepB/Hib Group (N=240) | Hiberix Group and Tritanrix-HepB Group (N=120)
Pain (General disorders) | 209/238 | 105/119
Redness (General disorders) | 128/238 | 76/119
Swelling (General disorders) | 166/238 | 83/119
Drowsiness (General disorders) | 73/238 | 34/119
Fever (General disorders) | 182/238 | 85/119
Irritability (General disorders) | 178/238 | 88/119
Loss of appetite (General disorders) | 96/238 | 49/119
Rhinitis (Infections and infestations) | 13 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.